CLINICAL TRIAL: NCT05872399
Title: Investigation of Greek Physiotherapy Students' Attitudes Towards Psychiatry and Mental Health
Brief Title: Greek Physiotherapy Students' Attitudes Towards Psychiatry and Mental Health
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Georgios Marios Kyriakatis, Undergraduate Student, Department of Physiothrapy, School of Health Sciences, University of Thessaly
Other Study IDs: 535, 2/5/2023
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Students; Physical Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physiotherapy students: The group will consist of Greek physiotherapy undergraduate students.
  Interventions: Other: Attitudes Towards Psychiatry - 30

INTERVENTIONS:
Other: Attitudes Towards Psychiatry - 30 — The participants will answer their beliefs in 30 statements about psychiatry and mental health.

SUMMARY:
The main purpose of this study will be to investigate what are the attitudes of Greek physiotherapy students who belong to one of the Higher Educational Institutions of Greece and the correlation of these attitudes with certain demographic characteristics that will be defined.

DETAILED DESCRIPTION:
A link will be created via google forms, which will be made available to undergraduate physiotherapy students of all the departments of the country's universities. The Attitudes Towards Psychiatry - 30 scale will be used to explore students' attitudes towards psychiatry and mental health. Participants through a mandatory field will consent to participate in the study, having read all the necessary information at the beginning. Then the necessary section will be created in which the participant will answer the questions of the assessment scale. The Attitudes Towards Psychiatry - 30 scale has not been standardized in Greek and for this reason it will be translated forward and backward by 2 independent researchers. After the completion of the study, the researchers will collect the results and draw conclusions based on the necessary statistical analyses. The data collection will be done for about one month, the duration of data processing and archiving will be about 6 months.

ELIGIBILITY:
Inclusion Criteria:

* physiotherapy student in one of the Universities of Greece

Exclusion Criteria:

* not a physiotherapy student at one of the country's Universities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include physiotherapy students that will have the ability of completing the assessment form.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Attitudes Towards Psychiatry - 30 | Only one time, at baseline.
  The scale will be completed by the participants themselves.

CONTACTS AND LOCATIONS:
Overall Officials: Phoebe Speis, Dr., Study Director — Αcademic fellow
Locations (1):
- University of Thessaly, Lamia, Fthiotis, Greece

REFERENCES:
- [Background] Connaughton J, Gibson W. Physiotherapy Students' Attitudes toward Psychiatry and Mental Health: A Cross-Sectional Study. Physiother Can. 2016;68(2):172-178. doi: 10.3138/ptc.2015-18E. PMID 27909364
- [Background] Probst M, Peuskens J. Attitudes of Flemish physiotherapy students towards mental health and psychiatry. Physiotherapy. 2010 Mar;96(1):44-51. doi: 10.1016/j.physio.2009.08.006. Epub 2009 Oct 24. PMID 20113762